CLINICAL TRIAL: NCT00279305
Title: Effects of Rituximab on the Progression of Type 1 Diabetes in New Onset Subjects
Brief Title: Rituximab in New Onset Type 1 Diabetes
Acronym: TN05
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); American Diabetes Association (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TN05 Ritux; U01DK061055 (NIH)
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Newly diagnosed type 1 diabetes; New Onset type 1 diabetes; Preservation of insulin secretion; Type 1 diabetes; Juvenile Onset Diabetes; Insulin Dependent Diabetes; T1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab Intravenous Infusion (Experimental): Participants will receive active rituximab (anti-CD20 monoclonal antibody) as an intravenous infusion, with 4 administrations at weeks 0, 1, 2, and 3 at a dose of 375mg/m2
  Interventions: Drug: Anti-CD20 (rituximab)
- Placebo Intravenous Infusion (Placebo Comparator): Participants will receive placebo given as an intravenous infusion with 4 administrations at weeks 0, 1, 2, and 3.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Anti-CD20 (rituximab)
  Arms: Rituximab Intravenous Infusion
Drug: Placebo Comparator — Placebo intravenous infusion
  Arms: Placebo Intravenous Infusion

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the immune system mistakenly attacks the insulin-producing beta cells in the pancreas. Without these beta cells, the body cannot maintain proper blood glucose levels in response to daily activities such as eating or exercise. With fewer insulin producing cells blood glucose increases, causing hunger, thirst, and unexplained weight loss. By the time these symptoms develop, 80-90% of a person's beta cells have already been destroyed. However, this also means that between 10-20% of these cells remain that continue to produce insulin.

Scientists have learned that two types of immune cells, B cells and T cells, are involved in causing type 1 diabetes. T cells are responsible for attacking and destroying the beta cells that make insulin. Although they don't attack insulin producing cells, B cells may be what trigger the T cells to attack.

This study will investigate the use of rituximab to see if it can help lower the number of immune B cells thereby preventing the destruction of any remaining insulin producing beta cells that remain at diagnosis. Rituximab is approved by the Food and Drug Administration (FDA) for the treatment of a condition called B-lymphocyte lymphoma. Its effects on the immune system are well understood through its use in organ transplantation. Research has shown that rituximab might be helpful in treating other conditions caused by T cells and B cells, including type 1 diabetes. The goal of this study is to find out if rituximab can preserve residual insulin secretion and prevent further beta cell destruction in type 1 diabetes.

DETAILED DESCRIPTION:
The study is a randomized, two-arm, trial in which 2/3 of participants will receive the study drug, while the remaining 1/3 will receive a placebo (a pretend medicine that does nothing). The group you are assigned to is decided by chance (as by the toss of a coin or drawing straws). Neither you nor your doctor will be able to choose which group you are in. Also, neither you nor the researchers will know which group you are in. Participants will take rituximab, or the placebo, once a week during the first 4 weeks in the study. It will be given as an intravenous infusion at a clinical center.

Participants will need to return to the clinical center for a visit about every 3 months for two years; those participants that continue to secrete insulin will have further follow-up for an additional two years.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 8 and 45 years
* Within 3 months of diagnosis of type 1 diabetes
* Have presence of at least one diabetes-related autoantibody
* Must have stimulated C-peptide levels of at least 0.2 pmol/ml measured during a mixed meal tolerance test (MMTT) within one month of randomization
* If female with reproductive potential, willing to avoid pregnancy and undergo pregnancy testing while participating in the study
* Have not received an immunization for at least one month
* Must be willing to comply with intensive diabetes management
* Must weigh at least 25 kg at study entry

Exclusion Criteria:

* Are immunodeficient or have clinically significant chronic lymphopenia
* Have an active infection or positive purified protein derivative (PPD) test result
* Currently pregnant or lactating; or anticipate becoming pregnant.
* Require chronic use of steroids
* Have current or past HIV, hepatitis B, or hepatitis C infection
* Have any complicating medical issues that interfere with study conduct or cause increased risk
* Have a history of malignancies
* Currently using non-insulin pharmaceuticals that effect glycemic control
* Currently participating in another type 1 diabetes treatment study

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Study Chair — Type 1 Diabetes TrialNet
Locations (16):
- United States (13):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California-San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Indiana University-Riley Hospital for Children, Indianapolis, Indiana
  - Joslin, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington
- Walter and Eliza Hall Institute of Medical Research, Victoria, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/tn05-anticd20/?query=tn05
URL: https://repository.niddk.nih.gov/studies/tn05-anticd20/?query=tn05

REFERENCES:
- [Background] Pescovitz MD. The use of rituximab, anti-CD20 monoclonal antibody, in pediatric transplantation. Pediatr Transplant. 2004 Feb;8(1):9-21. doi: 10.1046/j.1397-3142.2003.00135.x. PMID 15009836
- [Background] Noorchashm H, Noorchashm N, Kern J, Rostami SY, Barker CF, Naji A. B-cells are required for the initiation of insulitis and sialitis in nonobese diabetic mice. Diabetes. 1997 Jun;46(6):941-6. doi: 10.2337/diab.46.6.941. PMID 9166663
- [Background] Zecca M, Nobili B, Ramenghi U, Perrotta S, Amendola G, Rosito P, Jankovic M, Pierani P, De Stefano P, Bonora MR, Locatelli F. Rituximab for the treatment of refractory autoimmune hemolytic anemia in children. Blood. 2003 May 15;101(10):3857-61. doi: 10.1182/blood-2002-11-3547. Epub 2003 Jan 16. PMID 12531800
- [Background] Binstadt BA, Caldas AM, Turvey SE, Stone KD, Weinstein HJ, Jackson J, Fuhlbrigge RC, Sundel RP. Rituximab therapy for multisystem autoimmune diseases in pediatric patients. J Pediatr. 2003 Nov;143(5):598-604. doi: 10.1067/s0022-3476(03)00382-2. PMID 14615729
- [Background] Edwards JC, Leandro MJ, Cambridge G. B lymphocyte depletion in rheumatoid arthritis: targeting of CD20. Curr Dir Autoimmun. 2005;8:175-92. doi: 10.1159/000082103. PMID 15564721
- [Background] Sidner RA, Book BK, Agarwal A, Bearden CM, Vieira CA, Pescovitz MD. In vivo human B-cell subset recovery after in vivo depletion with rituximab, anti-human CD20 monoclonal antibody. Hum Antibodies. 2004;13(3):55-62. PMID 15598985
- [Background] Bearden CM, Agarwal A, Book BK, Vieira CA, Sidner RA, Ochs HD, Young M, Pescovitz MD. Rituximab inhibits the in vivo primary and secondary antibody response to a neoantigen, bacteriophage phiX174. Am J Transplant. 2005 Jan;5(1):50-7. doi: 10.1111/j.1600-6143.2003.00646.x. PMID 15636611
- [Background] Edwards JC, Szczepanski L, Szechinski J, Filipowicz-Sosnowska A, Emery P, Close DR, Stevens RM, Shaw T. Efficacy of B-cell-targeted therapy with rituximab in patients with rheumatoid arthritis. N Engl J Med. 2004 Jun 17;350(25):2572-81. doi: 10.1056/NEJMoa032534. PMID 15201414
- [Background] Serreze DV, Silveira PA. The role of B lymphocytes as key antigen-presenting cells in the development of T cell-mediated autoimmune type 1 diabetes. Curr Dir Autoimmun. 2003;6:212-27. doi: 10.1159/000066863. No abstract available. PMID 12408054
- [Result] Pescovitz MD, Greenbaum CJ, Krause-Steinrauf H, Becker DJ, Gitelman SE, Goland R, Gottlieb PA, Marks JB, McGee PF, Moran AM, Raskin P, Rodriguez H, Schatz DA, Wherrett D, Wilson DM, Lachin JM, Skyler JS; Type 1 Diabetes TrialNet Anti-CD20 Study Group. Rituximab, B-lymphocyte depletion, and preservation of beta-cell function. N Engl J Med. 2009 Nov 26;361(22):2143-52. doi: 10.1056/NEJMoa0904452. PMID 19940299
- [Derived] Pescovitz MD, Greenbaum CJ, Bundy B, Becker DJ, Gitelman SE, Goland R, Gottlieb PA, Marks JB, Moran A, Raskin P, Rodriguez H, Schatz DA, Wherrett DK, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet Anti-CD20 Study Group. B-lymphocyte depletion with rituximab and beta-cell function: two-year results. Diabetes Care. 2014 Feb;37(2):453-9. doi: 10.2337/dc13-0626. Epub 2013 Sep 11. PMID 24026563
- See also: Type 1 Diabetes TrialNet — http://www.diabetestrialnet.org
- See also: American Diabetes Association — http://www.diabetes.org
- See also: Juvenile Diabetes Foundation International — http://www.jdrf.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with newly diagnosed type 1 diabetes recruited from 12 TrialNet Clinical Centers between
Pre-assignment Details: 126 patients were assessed; 39 were excluded; 87 underwent randomization (57 were assigned to receive rituximab and 30 were assigned to receive placebo)
Groups:
- Rituximab Treatment: Four intravenous infusions (375 mg per square meter of body-surface area) were given on days 1, 8, 15, and 22 of the study
- Placebo: Placebo infusions were given to participants in control group on days 1, 8, 15, and 22.
Period: Overall Study
Arm/Group | Rituximab Treatment | Placebo
Started | 57 | 30
Completed | 49 | 29
Not Completed | 8 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Dificulting establishing IV | 1 | 0
Not completed — FDA Safety Alert | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab Treatment | Placebo | Total
Number analyzed (Participants) | 57 | 30 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.0 (8.6) | 17.4 (8.0) | 18.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 12 | 33
  Male | 36 | 18 | 54

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Stimulated C-peptide Curve Over the First 2 Hours of a 4-hour Mixed Meal Tolerance Test (MMTT) Administered at 1 Year
Description: The primary outcome is the area under the stimulated C-peptide curve (AUC) based on data collected at time 0 to 2 hours of a 4-hour mixed meal glucose tolerance test (MMTT) conducted at the primary endpoint visit. The timed measurements are done at: 0, 15, 30 60, 90, and 120 minutes.
  The calculation for the concentration of c-peptide is a weighted average of the 6 timed measurements of c-peptide in nano-moles/Liter. We try to distinguish this calculation from the AUC by referring to it as the "AUC mean" and may be expressed algebraically as the AUC/(120 min.); thus, the units are the same as the y-axis.
Time Frame: When all participants complete the 1 year visit
Measure: Mean (95% Confidence Interval); unit: pmol per mL
Arm/Group | Rituximab Treatment | Placebo
Number analyzed (Participants) | 49 | 29
pmol per mL | 0.58 [0.476 to 0.691] | 0.429 [0.289 to 0.585]
Statistical Analysis 1: Comparison: Rituximab Treatment vs Placebo; The calculation for the concentration of c-peptide is a weighted average of the 6 timed measurements of c-peptide in nano-moles/Liter. We try to distinguish this calculation from the AUC by referring to it as the "AUC mean" and may be expressed algebraically as the AUC/(120 min.); thus, the units are the same as the y-axis; Test type: Superiority or Other; p = 0.05, ANCOVA; Mean Difference (Final Values) = 0.139, 95% CI 2-sided [-0.0699 to 0.348], Standard Error of Mean 0.104

ADVERSE EVENTS:
Arm/Group | Rituximab Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 11/57 | 9/30
Other Adverse Events (participants affected / at risk) | 56/57 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Treatment (N=57) | Placebo (N=30)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (4) | 1 (2)
Sudden Death (General disorders) | 0 (0) | 1 (1)
Dermatology/Skin Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Endocrine- other (Endocrine disorders) | 2 (2) | 2 (3)
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 0 (0) | 1 (1)
Gastrointestinal Other (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection Other (Infections and infestations) | 0 (0) | 2 (2)
Infection with unknown ANC- pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC- Sinus (Infections and infestations) | 1 (1) | 0 (0)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Intra-operative Injury - Other (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Treatment (N=57) | Placebo (N=30)
Allergic rhinitis (Immune system disorders) | 10 (11) | 3 (5)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 0 (0) | 3 (9)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 7 (12) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 5 (7) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 11 (18) | 9 (14)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 12 (13) | 0 (0)
Vasovagal episode (Cardiac disorders) | 3 (5) | 2 (2)
Hypertension (Cardiac disorders) | 6 (6) | 0 (0)
Hypotension (Cardiac disorders) | 18 (25) | 5 (9)
Constitutional Symptoms - Other (General disorders) | 3 (3) | 2 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (8) | 2 (2)
Fever (General disorders) | 17 (19) | 5 (7)
Rigors/chills (General disorders) | 3 (3) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 6 (9) | 6 (7)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 21 (22) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 24 (26) | 3 (4)
Endocrine - Other (Endocrine disorders) | 0 (0) | 5 (5)
Dental: teeth (Gastrointestinal disorders) | 5 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 12 (15) | 3 (5)
Gastrointestinal - Other (Gastrointestinal disorders) | 4 (4) | 5 (6)
Nausea (Gastrointestinal disorders) | 25 (26) | 2 (2)
Vomiting (Gastrointestinal disorders) | 16 (19) | 3 (3)
Infection - Other (Infections and infestations) | 14 (15) | 2 (2)
Pelvis Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 3 (3) | 2 (2)
Skin Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 4 (4) | 2 (2)
Pharynx Infection with unknown ANC (Infections and infestations) | 8 (14) | 4 (8)
Sinus Infection with unknown ANC (Infections and infestations) | 3 (3) | 2 (6)
Upper Airway Infection with unknown ANC (Infections and infestations) | 14 (25) | 12 (22)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Fracture (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (4)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 12 (15) | 7 (11)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Neurology - Other (Nervous system disorders) | 3 (4) | 0 (0)
Sinus Pain (General disorders) | 13 (22) | 7 (13)
Other AE (General disorders) | 5 (7) | 4 (6)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Sexual/Reproductive Function - Other (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Flu-like syndrome (General disorders) | 4 (5) | 2 (2)
Vascular - Other (Vascular disorders) | 3 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No